CLINICAL TRIAL: NCT06560424
Title: Cardiovascular and Metabolic Sciences Biorepository
Status: Recruiting | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Wilson Tang, Staff Physician, Principal Investigator, The Cleveland Clinic
Other Study IDs: 24-708
Record Dates: First submitted 2024-08-13; First posted 2024-08-19 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Cardiovascular Diseases; Metabolic Disease
Keywords: Biorepository
MeSH Terms: conditions — Cardiovascular Diseases; Metabolic Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Blood (plasma, serum, whole blood, and/or PBMCs), urine, stool, and/or heart tissue samples.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Personal History of Cardiovascular or Metabolic Diseases: Persons who have a diagnosis of a cardiovascular or metabolic disease. Examples of cardiovascular diseases are: heart failure, arrhythmias, high cholesterol, coronary artery disease, heart attack, and stroke. Examples of metabolic diseases are: diabetes, metabolic syndrome, and hemochromatosis.
- Family History of Cardiovascular or Metabolic Diseases: Persons without a personal diagnosis of any cardiovascular or metabolic disease but with a family history in a first-degree relative of one of those diseases.
- Healthy Controls: No personal or family (first-degree relative) history of cardiovascular or metabolic diseases.

SUMMARY:
The purpose of the Cardiovascular and Metabolic Sciences Biorepository is to collect and store information and biospecimens (blood, urine, stool, and heart tissue) from patients with and without cardiovascular and metabolic diseases to create a readily available biorepository of samples and related medical health information to expedite future research into the causes and consequences of cardiovascular and metabolic diseases.

DETAILED DESCRIPTION:
Heart disease is the leading cause of death in the United States and other vascular diseases, like stroke, and metabolic diseases, like diabetes, are consistently in the top ten causes of death (CDC, 2024). There is clearly a need for continuing research and innovation into improved diagnosis and treatment of these diseases.

The goal of this biorepository is to provide an easily accessible collection of samples for researchers to utilize. The biorepository will also serve as a place to store residual samples from other cardiovascular disease (CVD) studies for future use, to make the best use of these biospecimen resources.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to sign the informed consent document

Exclusion Criteria:

* Chronic anemia (hemoglobin consistently <9 g/L)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We will enroll persons with diagnosed cardiovascular or metabolic disease(s), persons with a family history of cardiovascular and/or metabolic disease(s), and persons without known cardiovascular or metabolic disease(s). The targeted number of participants to be enrolled is indefinite.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2024-09-18 (Actual); Primary Completion 2050-12-31 (Estimated); Study Completion 2050-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of samples enrolled per year | Yearly through study completion (approximately 30 years)
  Establish a biorepository of samples (blood, urine, stool, and heart tissue) and related medical health information to support future investigation into cardiovascular and metabolic diseases.

CONTACTS AND LOCATIONS:
Overall Officials: W. H. Wilson Tang, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Main Campus, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided